CLINICAL TRIAL: NCT01193764
Title: Double Blind Placebo Controlled Study Assessing the Effect of Chocolate Consumption in Subjects With A History of Acne Vulgaris
Brief Title: Study Assessing the Effect of Chocolate Consumption in Subjects With A History of Acne Vulgaris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 20100520
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Acne
Keywords: acne; cocoa; chocolate; gelatin; pustule; comedones; papules; pustules
MeSH Terms: conditions — Acne Vulgaris | interventions — Chocolate; RID; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cocoa (Experimental): unsweetened 100% cocoa (Ghirardelli)
  Interventions: Dietary Supplement: 100% cocoa powder
- placebo (Placebo Comparator): hydrolyzed gelatin powder (Gelita)
  Interventions: Dietary Supplement: gelatin (Gelita)

INTERVENTIONS:
Dietary Supplement: 100% cocoa powder — A single-center, prospective, double blind, placebo controlled study will be conducted in which male subjects with very mild acne swallow capsules filled with either unsweetened 100% cocoa (Ghirardelli), hydrolyzed gelatin powder (Gelita), or a combination of the two, at baseline. The study team will fill the capsules with either 6 oz. of hydrolyzed gelatin, 6 oz. cocoa powder (Ghirardelli ©), or a 6 oz. combination of cocoa powder (Ghirardelli ©) and hydrolyzed gelatin, totaling 6oz using a capsule encapsulation sheet (holding 60 capsules that need to be filled each time). All subjects will ingest the same number of total capsules. Evaluations will be performed using clinical assessments 4 days and 7 days after baseline evaluations (+/- 1 days).
  Other Names: 100% cocoa powder (Ghirardelli ©); blue and white gelatin capsules (Capsuline)
  Arms: cocoa
Dietary Supplement: gelatin (Gelita) — A single-center, prospective, double blind, placebo controlled study will be conducted in which male subjects with very mild acne swallow capsules filled with either unsweetened 100% cocoa (Ghirardelli), hydrolyzed gelatin powder (Gelita), or a combination of the two, at baseline. The study team will fill the capsules with either 6 oz. of hydrolyzed gelatin, 6 oz. cocoa powder (Ghirardelli ©), or a 6 oz. combination of cocoa powder (Ghirardelli ©) and hydrolyzed gelatin, totaling 6oz using a capsule encapsulation sheet (holding 60 capsules that need to be filled each time). All subjects will ingest the same number of total capsules. Evaluations will be performed using clinical assessments 4 days and 7 days after baseline evaluations (+/- 1 days).
  Other Names: hydrolyzed gelatin (Gelita); blue and white gelatin capsules (Capsuline)
  Arms: placebo

SUMMARY:
The investigators conducted a recent pilot study and found a strong positive correlation between the consumption of 100% chocolate and acne exacerbation. However, this study had limitations including the lack of placebo and the small sample size. Although studies have been conducted assessing chocolate's effect on acne, no study has been done evaluating this effect using chocolate with 100% cocoa content in a double blind placebo controlled fashion. This study will analyze the difference in the number and type of acneiform lesions per subject at the different time points (Day 4 and Day 7) compared to baseline in order to increase the validity of the investigators results. In addition, the investigators will use unsweetened cocoa powder,12 rather than chocolate candy, which contains higher quantities of additive ingredients such as sugar and milk to avoid interference with the results and the possibility to establish or not an association between the unsweetened cocoa and an effect on acne.

ELIGIBILITY:
Inclusion Criteria:

* Post-pubescent males between the ages of 18-35 with minimal facial acne lesions defined as no less than 1 comedone and/or papule and no more than 8 total comedones and papules at Screening/Baseline
* Subjects who have no more than 2 papules at baseline
* Subjects who have no facial pustules at Screening/Baseline
* Subjects who have a history of facial acne vulgaris
* Subjects with a score of 0 or 1 on the investigator's Global Assessment Scale (See Appendix A)
* Subjects must sign an informed consent form
* Subjects must remain in the South Florida area during the study
* Volunteers in general good health
* Volunteers on no over the counter or prescribed medication, including supplements
* Subjects must be literate in the English language

Exclusion Criteria:

* Subjects of the female gender
* Subjects with a history of diabetes mellitus
* Subjects who have had allergic reactions to cocoa or gelatin
* Subjects who have more than 8 total comedones and papules at Screening/Baseline
* Subjects who have more than 2 papules at screening/baseline
* Subjects who have one or more pustules and/or nodules at Screening/Baseline
* Subjects with a history of taking anti-acne oral medication (i.e. isotretinoine) during the past six months
* Subjects who have used any oral antibiotics in the past two weeks
* Subjects currently applying any over-the-counter or prescribed anti-acne medication including, but not limited to, retinoic acid or benzoyl peroxide over the past six weeks
* Subjects who have used facial topical or injectable steroids 6 weeks prior to screening/baseline and during the study
* Subjects currently taking any over-the-counter or prescribed medication including but not limited to oral supplements, vitamin A, etc. over the past two weeks
* Subjects who used systemic corticosteroids 6 weeks prior to screening/baseline or during the study
* Subjects taking drugs known to be photosensitizers including, but not limited to, phenothiazines, amiodarone, quinine, thiazides, tetracyclines, sulphonamides, quinolones
* Subjects who are expected to have excess sun exposure during the study
* Subjects who will not be in the South Florida area during the study
* Subjects who are diagnosed with obesity with a BMI of 30 or greater
* Subjects who have a history of hypertriglyceridemia

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of acneiform lesions | 7 days
  Number of lesions counted.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Block, B.S., Study Director — University of Miami; Brian Berman, M.D., Ph.D., Principal Investigator — University of Miami; Caroline Caperton, M.D., M.S.P.H., Study Chair — University of Miami; Whitney Valins, B.S., Study Chair — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States